CLINICAL TRIAL: NCT04210206
Title: Kurzfristiger Einfluss Einer Guten Stoffwechseleinstellung Auf Kognitive Funktion, Wohlbefinden Und Stoffwechselparameter Bei Erwachsenen Patienten Mit Phenylketonurie (Short-term Effects of Good Metabolic Control on Cognitive Function, Wellbeing, and Metabolic Parameters in Adult Patients With Phenylketonuria)
Brief Title: Short-term Effects of Good Metabolic Control on Cognitive Function, Wellbeing, and Metabolic Parameters in Adult Patients With Phenylketonuria
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Klaus Parhofer (Other)
Responsible Party: Sponsor-Investigator, Klaus Parhofer, Professor of Endocrinology and Metabolism, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CoFu-PKU
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Phenylketonurias
Keywords: cognitive function adults
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet (Experimental)
  Interventions: Other: PHE-diet
- Control (No Intervention)

INTERVENTIONS:
Other: PHE-diet — phenylalanine-restricted diet with phenylalanine free supplements for 8 weeks
  Arms: Diet

SUMMARY:
The goal of this study is to evaluate if in adult patients with phenylketonuria (PKU) without strict metabolic control during the last 12 months, strict metabolic control for 8 weeks results in an improvement of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with classical PKU
* Age ≥ 18 years
* Good metabolic control during childhood (at least until 12 years of age)
* Plasma Phe levels ≥ 15 mg/dl for ≥ 1 year
* Written informed consent prior to study participation

Exclusion Criteria:

* Reduced cognitive function (unability to perform test battery)
* Drug and or alcohol abuse
* Treatment with BH4
* Treatment with drugs known to affect cognitive function

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Spatial working memory strategy index | 8 weeks
  cognitive function; scores range from 4 to 28, with lower scores representing better outcome

SECONDARY OUTCOMES:
Reaction time | 8 weeks
  cognitive function; milliseconds, with faster times representing better outcome
Paired Associates Learning | 8 weeks
  cognitive function; scores range from 0 to 70, with lower scores indicating better outcome
Multitasking Test | 8 weeks
  cognitive function; scores range from 0 to 279, with lower scores indicating better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University Munich, Munich, Germany